CLINICAL TRIAL: NCT05588908
Title: A Phase Ib/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection in Chinese Participants With Acute Gout
Brief Title: A Phase Ib/II Study of Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection in Chinese Participants With Acute Gout
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSGJ-613-AG-Ib/II-01
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Acute Gout
MeSH Terms: interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SSGJ-613 100 mg (phase Ib) (Experimental): Dose Arm 1 (phase Ib): SSGJ-613 100 mg subcutaneous (s.c) once. The s.c. injection could be administered into the abdomen or thigh.
  Interventions: Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 100 mg (phase Ib)
- SSGJ-613 200 mg (phase Ib) (Experimental): Dose Arm 2 (phase Ib): SSGJ-613 200 mg subcutaneous (s.c) once. The s.c. injection could be administered into the abdomen or thigh.
  Interventions: Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 200 mg (phase Ib)
- SSGJ-613 300 mg (phase Ib) (Experimental): Dose Arm 3 (phase Ib): SSGJ-613 300 mg subcutaneous (s.c) once. The s.c. injection could be administered into the abdomen or thigh.
  Interventions: Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 300 mg (phase Ib)
- SSGJ-613 200 mg (phase II) (Experimental): Dose Arm 4 (phase II): SSGJ-613 200 mg subcutaneous (s.c) once. The s.c. injection could be administered into the abdomen or thigh. Randomized patients will receive one s.c. injection of SSGJ-613 and placebo matching compound betamethasone injection (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection is recommended to be administered deeply into the gluteal muscle.
  Interventions: Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 200 mg (phase II)
- SSGJ-613 300 mg (phase II) (Experimental): Dose Arm 5 (phase II): SSGJ-613 300 mg subcutaneous (s.c) once. The s.c. injection could be administered into the abdomen or thigh. Randomized patients will receive one s.c. injection of SSGJ-613 and placebo matching compound betamethasone injection (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection is recommended to be administered deeply into the gluteal muscle.
  Interventions: Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection low dose 300 mg (phase II)
- Compound Betamethasone Injection 1 mL (phase II) (Active Comparator): Dose Arm 6 (phase II): Compound betamethasone injection 1 mL intramuscularly (i.m) once. The i.m. injection is recommended to be administered deeply into the gluteal muscle. Randomized patients will receive compound betamethasone injection 1 mL i.m. once and placebo matching SSGJ-613 s.c. once, on Day 1.
  Interventions: Drug: Compound Betamethasone Injection (phase II); Other: Placebo (phase II)

INTERVENTIONS:
Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 100 mg (phase Ib) — 100 mg subcutaneous (s.c) once
  Other Names: SSGJ-613 100 mg (phase Ib)
  Arms: SSGJ-613 100 mg (phase Ib)
Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 200 mg (phase Ib) — 200 mg subcutaneous (s.c) once
  Other Names: SSGJ-613 200 mg (phase Ib)
  Arms: SSGJ-613 200 mg (phase Ib)
Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 300 mg (phase Ib) — 300 mg subcutaneous (s.c) once
  Other Names: SSGJ-613 300 mg (phase Ib)
  Arms: SSGJ-613 300 mg (phase Ib)
Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 200 mg (phase II) — one s.c. injection of SSGJ-613 once, on Day 1.
  Other Names: SSGJ-613 200 mg (phase II)
  Arms: SSGJ-613 200 mg (phase II)
Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection low dose 300 mg (phase II) — one s.c. injection of SSGJ-613 once, on Day 1.
  Other Names: SSGJ-613 300 mg (phase II)
  Arms: SSGJ-613 300 mg (phase II)
Drug: Compound Betamethasone Injection (phase II) — 1 mL i.m. once on Day 1
  Arms: Compound Betamethasone Injection 1 mL (phase II)
Other: Placebo (phase II) — Participants will receive Placebo matching SSGJ-613 to maintain the blinding of the Investigational Medicinal Products.
  Other Names: PBO
  Arms: Compound Betamethasone Injection 1 mL (phase II)

SUMMARY:
The purpose of this study is to determine the target dose of phase II and to evaluate the safety, tolerability, pharmacokinetics and efficacy of recombinant anti-IL-1β humanized monoclonal antibody injection at different doses in Chinese participants with acute gout.

DETAILED DESCRIPTION:
The phase Ib study is a multi-center, open label, dose escalation study examining the effect of recombinant anti-IL-1β humanized monoclonal antibody injection and to determine the target dose of phase II for the treatment of acute flare in Chinese gout patients in whom non-steroidal anti-inflammatory drugs (NSAIDs) and/or colchicine are contraindicated, are not tolerated, or do not provide an adequate response. There are 3 dose groups (100 mg、200 mg and 300 mg) in phase Ib and 10 participants in each group.

The phase II study is a dose-ranging, multi-center, randomized, double-blind, double-dummy, active-controlled, parallel-group study examining the effect of 2 dose regimens (200 mg and 300 mg, based on the outcome of phase Ib) of recombinant anti-IL-1β humanized monoclonal antibody injection versus compound betamethasone injection for the treatment of acute flare in Chinese gout patients in whom NSAIDs and/or colchicine are contraindicated, are not tolerated, or do not provide an adequate response. The phase II recommended dose of SSGJ-613 in subjects with acute gouty was determined according to the phase Ib interim analysis results.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 Years to 65 Years, both male and female
* Meeting the American College of Rheumatology (ACR) 2015 criteria for the classification of acute arthritis of primary gout.
* Presence of acute gout flare for no longer than 7 days
* Baseline pain intensity > or = to 50 mm on the 0-100 mm VAS
* Contraindicated for, intolerant or unresponsive to NSAIDs, colchicine or both

Exclusion Criteria:

* Secondary gout (such as gout caused by chemotherapy, transplant gout, etc.)
* Evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis
* Presence of severe renal function impairment
* Intolerance of subcutaneous and intramuscular injection
* Known presence or suspicion of active or recurrent bacterial, fungal or viral infection at the time of enrollment
* History of malignant tumor within 5 years before screening
* Live vaccinations within 3 months prior to the start of the study
* Use of forbidden therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From baseline through 24 weeks
  To investigate the safety characteristics.
Phase Ib: Incidence and Severity of Abnormalities in Vital Signs/Physical Examinations, Laboratory Examinations and Other Relevant Examinations | From baseline through 24 weeks
  To investigate the safety characteristics.
Phase II: The Change in Pain Intensity in the Target Joint From Baseline to 72 Hours Post Dose as Measured on a 0-100 mm Visual Analog Scale (VAS) | Baseline, at 72 hrs post-dose
  The change in pain intensity from baseline to 72 hours post dose as measured on a 0-100 mm Visual Analog Scale (VAS): 0= no pain and 100= severe pain. Change from baseline = (post-baseline measurement - baseline).

SECONDARY OUTCOMES:
Phase Ib: Pharmacokinetic (PK) Cmax | From baseline through 24 weeks
  PK parameters (Cmax) following single dose.
Phase Ib: Pharmacokinetic (PK) Tmax | From baseline through 24 weeks
  PK parameters (Tmax) following single dose.
Phase Ib: Pharmacokinetic (PK) AUC 0-t | From baseline through 24 weeks
  PK parameters (AUC 0-t) following single dose.
Phase Ib: Pharmacokinetic (PK) AUC 0-∞ | From baseline through 24 weeks
  PK parameters (AUC 0-∞) following single dose.
Phase Ib: Pharmacokinetic (PK) t1/2 | From baseline through 24 weeks
  PK parameters (t1/2) following single dose.
Phase Ib: The Pain Intensity in the Target Joint at 6, 12, 24, 48, 72 Hours, 4, 5, 6, 7 Days, and 4, 8, 12, 16, 20, 24 Weeks Post Dose as Measured on a 0-100 mm Visual Analog Scale (VAS) | At 6, 12, 24, 48, 72 Hours, 4, 5, 6, 7 Days, and 4, 8, 12, 16, 20, 24 Weeks post-dose
  The pain intensity post dose as measured on a 0-100 mm Visual Analog Scale (VAS): 0= no pain and 100= severe pain.
Phase II: The Pain Intensity in the Target Joint at 6, 12, 24, 48, 72 Hours, 4, 5, 6, 7 Days, and 4, 8, 12 Weeks Post Dose as Measured on a 0-100 mm Visual Analog Scale (VAS) | At 6, 12, 24, 48, 72 Hours, 4, 5, 6, 7 Days, and 4, 8, 12 Weeks post-dose
  The pain intensity post dose as measured on a 0-100 mm Visual Analog Scale (VAS): 0= no pain and 100= severe pain.
The Change in Pain Intensity in the Target Joint From Baseline to 6, 12, 24, 48 Hours Post Dose as Measured on a 0-100 mm Visual Analog Scale (VAS) | Baseline, at 6, 12, 24, 48 hrs post-dose
  The change in pain intensity from baseline to 6, 12, 24, 48 hours post dose as measured on a 0-100 mm Visual Analog Scale (VAS): 0= no pain and 100= severe pain. Change from baseline = (post-baseline measurement - baseline).
The Time to At Least 50% Reduction of Baseline Pain Intensity in the Target Joint Within 7 Days after study drug administration | Baseline, within 7 days after study drug administration
  The time to at least 50% reduction in Pain intensity from baseline as measured by Visual Analog Scale (VAS) for each treatment group, is estimated using the Kaplan Meier method. Participants scored their pain intensity in the target joint on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100).
The Time to Complete Pain Remission of Baseline Pain Intensity in the Target Joint Within 12 Weeks after study drug administration | Baseline, within 12 weeks after study drug administration
  The time to complete pain remission in Pain intensity from baseline as measured by a 5-point Likert scale for each treatment group, is estimated using the Kaplan Meier method. Participants scored their pain intensity in the target joint on a 5-point Likert scale: None, mild, moderate, severe, extremely severe.
Percentage of Participants Taking Rescue Medication Within 7 Days After Study Drug Administration | 7 days after study drug administration
  Participants who had difficulty in tolerating their pain after the 12 and 72 hours post-dose pain assessments were allowed to take rescue medication.

CONTACTS AND LOCATIONS:
Overall Officials: Hejian Zou, MD, Principal Investigator — Shanghai Huanshan Hospital Fudan University-Rheumatology; Qinghong Zhou, MD, Study Director — Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd.
Locations (3):
- China (3):
  - Site 02, Wuhan, Hubei
  - Site 03, Linyi, Shandong
  - Site 01, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No